CLINICAL TRIAL: NCT04445454
Title: Mesenchymal Stromal Cell Therapy for Severe Covid-19 Infection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Yves Beguin, MD,PhD, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJT2012
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Coronavirus Infection
Keywords: mesenchymal stromal cells
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: This study is a monocentric prospective phase I/II clinical trial, aiming at evaluating the safety and efficacy of 3 intravenous administrations of BM-MSC in 20 patients with severe to critical COVID-19 pneumonia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC therapy for severe COVID-19 infection (Experimental): After signed informed consent, patients will receive 3 infusions of (1.5)-3.0 x106/kg BM-MSC (from the same donor) at 3-4 days interval, in addition to the standard of care for COVID-19 disease.
  Interventions: Biological: Mesenchymal stromal cells

INTERVENTIONS:
Biological: Mesenchymal stromal cells — Bone marrow collection and MSC expansion cultures will be carried out at the Laboratory of Cell and Gene Therapy (LTCG) at the University of Liège as described in IMPD and its SOPs.
  Other Names: MSC

SUMMARY:
The overall objective of the study is to evaluate the safety and efficacy of MSC therapy combined with best supportive care in hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
This study is a monocentric prospective phase I/II clinical trial, aiming at evaluating the safety and efficacy of 3 intravenous administrations of BM-MSC in 20 patients with severe to critical COVID-19 pneumonia.

After signed informed consent, patients will receive 3 infusions of (1.5)-3.0 x106/kg BM-MSC (from the same donor) at 3-4 days interval, in addition to the standard of care for COVID-19 disease.

The trial will be open for inclusion for 2 years after initiation. Each patient will be followed for 90 days after inclusion. The total study duration will thus be 2 years and 90 days.

ELIGIBILITY:
COVID-19 patients Inclusion criteria

* Male or female patients aged at least 18 years and up to 70 years
* Diagnosed with microbiologically or radiologically confirmed COVID-19 pneumonia as defined by:
* Extensive interstitial pneumonia on CT scan, consistent with viral pneumonia, within 10 days prior to randomization
* And either positive result of COVID-19 PCR test within 14 days prior to inclusion or positive result of SARS-CoV2 PCR or serology within 14 days after inclusion.
* Requiring oxygen administration (SpO2 ≤ 93% on room air):

  * Group A: in standard or intensive care unit requiring supplemental oxygen
  * Group B: in intensive care unit under mechanical ventilation administered through a tracheal tube, either:
* for less than or equal to 7 days
* for 7 to 14 days, with persisting high inflammation (ferritin > 2,000 µg/L; ferritin > 1,000 µg/L and rising; lymphocytes < 800 with CRP > 70 mg/L and rising or ferritin > 700 µg/L and rising or LDH > 300 UI/L or D-Dimers > 1000 ng/ml), not explained by superinfection. Rising = compared to previous 24H.
* Written consent of the patient, or - if impossible (clinical condition precluding capacity to consent) - of his/her legal representative, or - if impossible - of an impartial witness such as a physician from a non-participating department or member of the Ethics Committee. Any consent obtained this way shall be documented and confirmed by way of normal consent procedures at the earliest opportunity when the patient has recovered

Exclusion criteria

* Ongoing pregnancy. Women of childbearing potential (WOCBP, defined as a premenopausal female capable of becoming pregnant) should use an appropriate method of contraception (oral, injectable, or mechanical contraception; women whose partners have been vasectomized or have received or are utilizing mechanical contraceptive devices).
* Extracorporeal membrane oxygenation
* Limitations to intensity of care
* Life expectancy < 24 hours
* Known allergy to IMP component
* Active secondary infection
* Any malignancy (except non-melanoma skin carcinoma) within 2 years before inclusion
* Pre-existing thrombo-embolic pathology
* Signs of an active drug or alcohol dependence, serious current illness, mental illness or any factors which, in the opinion of the Investigator, may interfere with subject's ability to understand and comply with study requirements
* Patients with any serious medical condition or abnormality of clinical laboratory tests that, in the Investigator's judgment, precludes the patient's safe participation in and completion of the study.
* Participation in another clinical trial(use of anti-viral/supportive drugs for COVID-19 infection on a compassionate use basis is not an exclusion criterion).

MSC donors Inclusion criteria

* Unrelated to the patient
* Male or female
* Age > 18 yrs
* No HLA matching required
* Fulfills generally accepted criteria for allogeneic HSC donation
* Informed consent given by donor

Exclusion criteria

* Any condition not fulfilling inclusion criteria
* Known allergy to lidocaine
* Any risk factor for transmissible infectious diseases, in particular HIV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of intravenous infusion of MSC in patients with severe to critical COVID-19 pneumonia | Day 28
  To assess the infusional toxicity
To evaluate the safety of intravenous infusion of MSC in patients with severe to critical COVID-19 pneumonia | Day 28
  To assess the number of Adverse events of special interest : Incidence of infections (bacterial, viral, fungal, parasitic) and thrombo-embolic events.
To evaluate the efficacy of intravenous infusion of MSC in patients with severe to critical COVID-19 pneumonia | Day 28
  Group A (patients not under mechanical ventilation): to determine the pourcentage of patients requiring mechanical ventilation
To evaluate the efficacy of intravenous infusion of MSC in patients with severe to critical COVID-19 pneumonia | Day 28
  Group B (patients under mechanical ventilation): to determine the vital status (dead/alive)

SECONDARY OUTCOMES:
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 28
  To assess the clinical status (on a 7-point WHO ordinal scale)
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 28
  To assess the duration of oxygen therapy and/or mechanical ventilation
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 90
  To assess the length of stay at the intensive care unit and of hospitalization
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 28
  To assess the number of organ failures
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 28
  To assess the intensity of the inflammatory response
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 28
  To assess the evolution of coagulation parameter
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 28
  To assess the presence of Biomarker of lung lesion, repair and scarring
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 90
  To assess the v iral load over the 28 days after inclusion and seroconversion to COVID-19 over the 90 days after inclusion
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 90
  To assess the pulmonary function
To evaluate the effect of MSC administration associated with the standard of care (SOC including anti-viral therapy) | Day 90
  To assess the number of adverse reactions (ARs), ARs grade > 3, serious adverse events (SAEs), serious ARs (SARs), suspected expected and unexpected SARs (SESARs and SUSARs).

OTHER OUTCOMES:
To investigate immune modulation | Day 28
  To determine the FACS analysis of regulatory T-cell (Treg) levels and Treg and Tconv sub-populations
To compare the cytotoxic activity of PBMCs from healthy control and COVID-19 patients (divided in responders / non-responders to MSC therapy) against MSCs in vitro | Day 28
  To assess the cytotoxic activity by MLR

CONTACTS AND LOCATIONS:
Overall Officials: Yves Beguin, MD,PhD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gregoire C, Layios N, Lambermont B, Lechanteur C, Briquet A, Bettonville V, Baudoux E, Thys M, Dardenne N, Misset B, Beguin Y. Bone Marrow-Derived Mesenchymal Stromal Cell Therapy in Severe COVID-19: Preliminary Results of a Phase I/II Clinical Trial. Front Immunol. 2022 Jul 4;13:932360. doi: 10.3389/fimmu.2022.932360. eCollection 2022. PMID 35860245